CLINICAL TRIAL: NCT00008151
Title: Gemtuzumab Ozogamicin (GO), Fludarabine, And Low-Dose TBI Followed By Donor Stem Cell Transplantation For Patients With Advanced Acute Myeloid Leukemia Or Myelodysplastic Syndrome
Brief Title: Gemtuzumab Ozogamicin, Fludarabine, and Total-body Irradiation Followed by Peripheral Stem Cell or Bone Marrow Transplantation in Treating Patients With Advanced Acute Myeloid Leukemia or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 1555.00; FHCRC-1555.00; NCI-G00-1900; CDR0000068383+ (Registry Identifier: PDQ)
Record Dates: First submitted 2001-01-06; First posted 2004-03-25 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-03

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts | interventions — Cyclosporine; fludarabine phosphate; Gemtuzumab; Methotrexate; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Drug: cyclosporine
Drug: fludarabine phosphate
Drug: gemtuzumab ozogamicin
Drug: methotrexate
Drug: mycophenolate mofetil
Procedure: allogeneic bone marrow transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Monoclonal antibodies such as gemtuzumab ozogamicin can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Peripheral stem cell or bone marrow transplantation may be able to replace immune cells that were destroyed by chemotherapy and radiation therapy used to kill cancer cells.

PURPOSE: Phase II trial to study the effectiveness of gemtuzumab ozogamicin combined with fludarabine and total-body irradiation followed by donor peripheral stem cell or bone marrow transplantation in treating patients who have advanced acute myeloid leukemia or myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response and disease-free survival at 1 year of patients with advanced acute myeloid leukemia or myelodysplastic syndrome treated with gemtuzumab ozogamicin, fludarabine, and total body irradiation followed by allogeneic peripheral blood stem cell or bone marrow transplantation with cyclosporine and mycophenolate mofetil. II. Determine the leukemic blast clearance from the blood and marrow in these patients treated with this regimen. III. Determine the safety and pharmacokinetics of gemtuzumab ozogamicin as part of this regimen in these patients. IV. Determine the incidence of donor stem cell engraftment in these patients. V. Determine the incidence and severity of graft-versus-host disease in these patients treated with this regimen. VI. Determine whether donor lymphocyte infusion can be safely used in the patients with mixed or full donor chimerism to eliminate persistent or progressive disease.

OUTLINE: Patients receive gemtuzumab ozogamicin IV over 2 hours on days -21 (first 5 patients) or -14 (subsequent patients) and -7, and fludarabine IV over 2 hours on days -4 to -2. Patients undergo total body irradiation followed by infusion of allogeneic peripheral blood stem cells or bone marrow on day 0. Patients receive oral or IV cyclosporine 2-3 times daily on days -3 to 56 (if related donor) or 100 (if unrelated donor) and oral or IV mycophenolate mofetil twice daily on days 0 to 27 (if related donor) or 40 (if unrelated donor). Patients receive 2 doses of intrathecal methotrexate prior to transplant and an additional 4 doses after transplant. Patients with cerebral spinal fluid (CSF) positive for malignant cells instead receive intrathecal cytarabine, methotrexate and hydrocortisone prior to transplant twice weekly until CSF blasts clear. Patients with persistent or recurrent disease after transplant may receive up to 3 donor lymphocyte infusions if graft-versus-host disease is less than grade II and they have greater than 5% donor CD3 cells. Patients are followed at 6 months and then annually thereafter.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study within 1-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of recurrent or refractory acute myeloid leukemia CD33 positive Greater than 5% morphologically identified blasts in the marrow OR Diagnosis of myelodysplastic syndrome CD33 positive Greater than 5% morphologically identified blasts in the marrow (refractory anemia with excess blasts (RAEB) and RAEB in transformation) Must have donor who meets the following criteria: HLA-A, B, C, DRB1 and DQB1 identical or mismatched for no more than 1 allelic or cross-reactive antigen Under 75 years of age

PATIENT CHARACTERISTICS: Age: Any age Performance status: Not specified Life expectancy: Not specified Hematopoietic: WBC no greater than 30,000/mm3 (leukophereses or hydroxyurea allowed) Hepatic: Bilirubin no greater than 2 times upper limit of normal No synthetic dysfunction No severe cirrhosis Renal: Not specified Cardiovascular: No symptomatic coronary artery disease No cardiac failure requiring therapy Pulmonary: DLCO at least 35% OR Receiving supplementary continuous oxygen Other: No uncontrolled infection No other diseases that would severely limit life expectancy Not pregnant or nursing Fertile patients must use effective contraception during and for 1 year after study

PRIOR CONCURRENT THERAPY: No post-transplant growth factors during and for 1 month after mycophenolate mofetil administration

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-10; Primary Completion 2002-07 (Actual); Study Completion 2002-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sievers, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States